CLINICAL TRIAL: NCT05504473
Title: Blink Restoration in Patients With Facial Nerve Palsy
Acronym: NEURO-BLINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Aarau (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Principal Investigator, Anthia Papazoglou, Prinicipal Investigator, Kantonsspital Aarau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB01
Record Dates: First submitted 2021-10-30; First posted 2022-08-17 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Facial Nerve Palsy
Keywords: neurostimulation; orbicularis oculi
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with facial nerve palsy and lagophthalmus (Experimental): There is only one arm in this study. The investigators examine if the medical device can achieve a painless blinking in patients with facial nerve palsy and lagophthalmus.
  Interventions: Device: NEURO-BLINK Device

INTERVENTIONS:
Device: NEURO-BLINK Device — The NEURO-BLINK is a class IIa medical device that intends to restore the blink function in patients with facial palsy through the application of transcutaneous electrical stimulation.

SUMMARY:
This study is a non-blinded single armed pilot study aiming to apply a newly created medical device in patients with seventh nerve palsy suffering from lagophthalmus in order to determine the best way for neuromuscular stimulation of the orbicularis oculi muscle and facial nerve in order to enable eyelid closure (blink). Initially, a tailored external neurostimulation prototype will be created in collaboration with the ETH for patients with facial nerve palsy and lagophthalmos. Aim of this study is to create an efficient, safe and comfortable medical device that can achieve an effective blinking through external electrical neuromuscular stimulation of the orbicularis oculi in patients with facial palsy and lagophthalmos. Such a device can become an essential part of facial palsy treatment.

DETAILED DESCRIPTION:
Facial paralysis rates are reported to be 4/10,000 per annum leading to facial asymmetry and impairs essential facial functions, including blinking, protection of the cornea, lip competence, mastication, speaking, but also has psychosocial penalties.

Facial animation is orchestrated by the facial muscles directed by the facial nucleus through a network of the facial nerve and its branches. The facial nerve (CNVII) plays a critical role in multiple complex functions of human life including mastication, speech, and successful social communication through expression of mood and emotion. The absence of facial nerve's function can be a result of a developmental anomaly, of a stroke leading to a damage to the central segment of this nerve (facial nucleus in the pons, motor cortex, or connections between the two), an iatrogenic or traumatic injury, a neoplastic infiltration or an infectious (e.g., borreliosis and herpes zoster), or idiopathic inflammation of the extratemporal segments of the facial nerve. The peripheral facial paralysis (PFP), resulting from affection of the seventh nerve is the most common pathology of the cranial pairs.

The facial nerve normally emits electrical impulses to give muscles their tone and shape. Therefore, when it is damaged, the muscles become weak and floppy. External electrical stimulation can mimic the electrical nerve impulses and help restore muscle tone in patients with facial palsy. Applications involving nerve stimulation can be divided into three separate categories: therapeutic electrical stimulation (TES), neuromodulatory stimulation (NMS), and functional electrical stimulation (FES). By FES standards, neural prosthetic reanimation of the eyelids for blink restoration is a relatively simple and low-risk application. Restoration of blinking involves a single muscle, the orbicularis oculi. The presence of the nerve is not required for external electrical stimulation to be used.

External electrical neuromuscular stimulation can try to mimic the electrical nerve impulses in patients with facial palsy. However, no device has yet been proven appropriate for daily use. The research question the investigators aim to answer is whether an efficient, safe and comfortable medical device that can achieve an effective blinking through external electrical neuromuscular stimulation of the orbicularis oculi in patients with facial palsy and lagophthalmos can be created. The stimulation will be provided in the form of charge balanced biphasic square pulses as shown in the image below at a frequency of 100Hz. The investigators mainly want to determine the functionality of a constant external electrostimulation for the patients. Blinking sufficiency will be evaluated qualitatively and quantitatively through surveys and observations.

The investigators aim to recruit initially 10 patients suffering from lagophthalmos due to facial nerve palsy, who will be invited to wear the device. The exact parameters needed for the neurostimulation and symptoms of patients or any adverse events will be documented on the case report form (CRF).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Facial palsy
* Lagophthalmus

Exclusion Criteria:

* Minors
* Pacemaker or defibrillator
* Vulnerable population
* Patients in emergency situations
* Allergies on the sticky electrodes and MD metallic sensors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
External electrical stimulation for a painless eye closure - Percentage of Eye closure (Parameter 1) | 2 year
  The investigators aim to use external electrical neuromuscular stimulation in order to achieve eye blinking/closure in 10 patients with lagophthalmos due to facial nerve palsy. In particular, the inverstigators aim to measure: Percentage of Eye closure during blink (between supported condition and pathological condition)
External electrical stimulation for a painless eye closure - Percentage of cornea coverage during blink (Parameter 2) | 2 year
  The investigators aim to use external electrical neuromuscular stimulation in order to achieve eye blinking/closure in 10 patients with lagophthalmos due to facial nerve palsy. In particular, we measure: Percentage of cornea coverage during blink (between supported condition and pathological condition) measured in mm
External electrical stimulation for a painless eye closure - Lagophthalmos reduction in mm (Parameter 3) | 2 year
  The investigators aim to use external electrical neuromuscular stimulation in order to achieve eye blinking/closure in 10 patients with lagophthalmos due to facial nerve palsy. In particular, the inverstigators measure: Lagophthalmos reduction during closed eyes (between supported condition and pathological condition) measured in mm
External electrical stimulation for a painless eye closure - Visual acuity (Parameter 4) | 2 year
  The investigators aim to use external electrical neuromuscular stimulation in order to achieve eye blinking/closure in 10 patients with lagophthalmos due to facial nerve palsy. In particular, the inverstigators measure: Visual acuity before and after the treatment through electronic Snellen charts
External electrical stimulation for a painless eye closure - influence upon corneal eye dryness (Parameter 5) | 2 year
  The investigators aim to use external electrical neuromuscular stimulation in order to achieve eye blinking/closure in 10 patients with lagophthalmos due to facial nerve palsy. In particular, the inverstigators measure: eye dryness before and after the treatment through Oxford scale
External electrical stimulation for a painless eye closure - influence upon quality of life in reference to eye dryness (Parameter 6) | 2 year
  The investigators aim to use external electrical neuromuscular stimulation in order to achieve eye blinking/closure in 10 patients with lagophthalmos due to facial nerve palsy. In particular, the inverstigators measure: dry eye questionnaire through OSDI and McGill quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Menke, Study Chair — Cantonal Hospital Aarau Ophthalmology Department
Locations (1):
- Ophthalmology Department Cantonal Hospital Aarau, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No